CLINICAL TRIAL: NCT04981236
Title: Pericapsular Nerve Group (PENG) Block Versus Periarticular Injection for Pain Management After Total Hip Arthroplasty: a Randomized Controlled Trial
Brief Title: Pericapsular Nerve Group (PENG) Block Versus Periarticular Injection for Pain Management After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2021-0725
Record Dates: First submitted 2021-07-22; First posted 2021-07-28 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Total Hip Arthroplasty; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group block (Active Comparator): Participants receiving pericapsular nerve group block
  Interventions: Procedure: Pericapsular nerve group block
- Periarticular block (Experimental): Participants receiving periarticular block
  Interventions: Procedure: Periarticular block

INTERVENTIONS:
Procedure: Pericapsular nerve group block — A curvilinear 2-5MHz ultrasound probe will be initially placed in a transverse plane over the anterior superior iliac spine and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the iliopubic eminence, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A 22-gauge, 80-mm needle will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. A total volume of 20 ml of ropivacaine 0.3% will be injected.
  Other Names: PENG block
  Arms: Pericapsular nerve group block
Procedure: Periarticular block — The periarticular injection solution contained 20mL of 7.5 mg/mL ropivacaine, 30mg of ketorolac, and 0.3mL of 1.0 mg/mL epinephrine. These agents were mixed with normal saline to a combined volume of 50mL. The surgeon injected this mixture into the tensor fascia lata, subcutaneous tissues, abductors, short external rotators muscles, and structures in the capsule.
  Arms: Periarticular block

SUMMARY:
Adequate pain control after total hip arthroplasty is crucial for early ambulation and patient satisfaction. The pericapsular nerve group (PENG) block has been recently introduced a new technique for blockade of the articular branches of the femoral, obturator and accessory obturator nerves. PENG block provides sufficient analgesia but it is still the potential for quadriceps weakness that might delay ambulation. Periarticular injection has attached attention as an effective analgesic modality with a low prevalence of adverse effects. The investigators will compare ultrasound-guided PENG block with periarticular injection in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 19 years old or older
2. American Society of Anesthesiologists Physical Status 1-3
3. Scheduled for elective unilateral total hip arthroplasty

Exclusion Criteria:

1. Allergy or intolerance to any of the drugs used in the study
2. Hepatic or renal insufficiency
3. Opioid dependency
4. Coagulopathy
5. Pre-existing neurologic or anatomic deficits in the lower extremities
6. Severe psychiatric illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale pain score | at 24 hours postoperatively
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) at 24 hours postoperatively

SECONDARY OUTCOMES:
Numeric rating scale pain score | at 6 hours postoperatively and 48h postoperatively
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) at 6 hours postoperatively and 48h postoperatively
Quadriceps muscle strength | at 24 hours postoperatively
  Quadriceps muscle strength will be measured by the dynamometer at 24h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Yong Seon Choi, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, Republic of Korea
Locations (1):
- Division of Cardiac Anesthesiology, Department of Anesthesiology and Pain Medicine, Cardiovascular Hospital, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No